CLINICAL TRIAL: NCT02142803
Title: A Phase 1 Study of MLN0128 and Bevacizumab in Patients With Recurrent Glioblastoma and Other Solid Tumors
Brief Title: TORC1/2 Inhibitor MLN0128 and Bevacizumab in Treating Patients With Recurrent Glioblastoma or Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01118; NCI-2014-01118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14-079; 9552 (Other: Dana-Farber Cancer Institute); 9552 (Other: CTEP); P30CA006516 (NIH); U01CA062490 (NIH); U01CA076576 (NIH); UM1CA186709 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-08

CONDITIONS: Adult Glioblastoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Malignant Uterine Corpus Neoplasm; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Solid Neoplasm; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Glioblastoma; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (TORC1/2 inhibitor INK128, bevacizumab) (Experimental): Patients receive TORC1/2 inhibitor INK128 PO QD on days 1-28 and bevacizumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sapanisertib

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sapanisertib — Given PO
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228

SUMMARY:
This phase I trial studies the side effects and best dose of raptor/rictor-mammalian target of rapamycin (mTOR) (TORC1/2) inhibitor MLN0128 when given in combination with bevacizumab in treating patients with glioblastoma, a type of brain tumor, or a solid tumor that has spread and not responded to standard treatment. TORC1/2 inhibitor MLN0128 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the progression of tumors by blocking the growth of new blood vessels necessary for tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose and recommended phase 2 dose (MTD/RP2D) of daily oral MLN0128 (TORC1/2 inhibitor INK128) when administered with bevacizumab in patients with advanced solid tumors including recurrent glioblastoma (GBM).

II. To evaluate the overall safety and tolerability of the combination of MLN0128 and bevacizumab.

SECONDARY OBJECTIVES:

I. To assess the preliminary anti-tumor activity of the combination of MLN0128 and bevacizumab, as determined by response rate (RR), progression-free survival (PFS) and overall survival (OS).

II. To assess tolerability throughout study therapy with MLN0128 and bevacizumab, including beyond the MTD interval with the following measures of cumulative treatment-related toxicities: frequency of toxicities leading to missed doses or delays; percentage of cycles given or not within 7 days of their scheduled times; percentage of actual planned dosage administration; percentage of patients that discontinue study drugs due to treatment related toxicity.

TERTIARY OBJECTIVES:

I. To assess cerebrospinal fluid (CSF) penetration of MLN0128 in combination with bevacizumab in patients with recurrent GBM by evaluating the plasma and CSF concentrations of MLN0128 in the absence and presence of bevacizumab.

II. To perform archival tumor analysis for markers of dysregulated cell signaling that may predict response to mechanistic target of rapamycin (mTOR) inhibitor therapy such as epidermal growth factor receptor (EGFR) (expression by immunohistochemistry [IHC] and amplification by fluorescent in situ hybridization [FISH]), phosphatase and tensin homolog (PTEN) (expression by IHC and deletion by FISH), phosphorylated (p)-protein kinase B (AKT), p-ribosomal protein S6 kinase (S6K), p-eukaryotic translation initiation factor 4E binding protein 1 (4EBP), p-mTOR and p-mitogen-activated protein kinase 1 (Erk) in patients with recurrent GBM.

III. To analyze select phosphorylated proteins (ERK, AKT, mTOR, 4EBP1, glycogen synthase kinase 3-beta [GSK3beta], ribosomal protein S6 kinase, 70kDa, polypeptide 2 [p70S6K], rS6) from tumor biopsies obtained at baseline and after treatment with MLN0128 from endometrial and ovarian cancer patients enrolled in stage 2.

IV. To analyze circulating plasma levels of angiogenic growth factors before, during and after treatment with MLN0128 and bevacizumab V. To perform genetic mutation analysis and proteomic analysis of tissue from biopsies of endometrial and ovarian cancer patients including analysis of Kirsten rat sarcoma viral oncogene homolog (KRAS), v-raf murine sarcoma viral oncogene homolog B (BRAF), phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA), v-akt murine thymoma viral oncogene homolog 1 (AKT1) and PTEN.

OUTLINE: This is a dose-escalation study of MLN0128.

Patients receive TORC1/2 inhibitor MLN0128 orally (PO) once daily (QD) and bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically/cytologically confirmed diagnosis of recurrent glioblastoma or an advanced solid tumor in which bevacizumab has shown benefit in specific disease population and for which standard or curative measures do not exist or are no longer effective
* Measurable or evaluable disease as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for non-GBM tumors and by Response Assessment in Neuro-Oncology (RANO) criteria for GBM
* For stage 1 (all patients) and dose expansion (stage 2) endometrial and ovarian cancer cohorts, participants are allowed following unlimited prior therapy; for stage 2 GBM participants, no more than 2 prior relapses are allowed; for these patients, relapse is defined as progression following initial therapy (i.e. radiation +/- chemo if that was used as initial therapy) or a subsequent therapy; the intent therefore is that GBM patients enrolling onto stage 2 had no more than 3 prior therapies (initial and treatment for 2 relapses); if the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered to constitute 1 relapse

  * NOTE: for participants who had prior therapy for a low-grade glioma, the surgical diagnosis of glioblastoma will be considered the first relapse; therefore, these participants may have had more than 3 prior therapies
* Patients must have recovered from clinically significant toxicity of prior therapy to grade =< 1 or pre-treatment baseline; the following intervals from previous treatments are required prior to day 1 of study therapy:

  * 12 weeks from the completion of radiation for recurrent GBM unless there is surgical diagnosis of recurrence or a new lesion that was not previously radiated
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from an investigational agent (not Food and Drug Administration [FDA] approved) (or 5 half lives, whichever is shorter)
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., erlotinib, hydroxychloroquine, etc.) (or 5 half lives, whichever is shorter)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin < 1.5 x institutional upper limit of normal with direct bilirubin within normal limits except for participants with Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (=< 5 x upper limit of normal [ULN] if liver metastases are present)
* Creatinine < 1.5 x normal institutional limits OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine level above institutional normal based either on Cockroft-Gault estimate or based on urine collection (12 or 24 hour)
* Metabolic: fasting serum glucose (=< 130 mg/dL) and fasting triglycerides =< 300 mg/dL
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 6 months after completion of MLN 0128 or bevacizumab administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of MLN0128 or bevacizumab administration
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= three years prior to registration
* Solid tumor patients must be off corticosteroids prior to registration; if GBM patient is receiving corticosteroids, patient must be on a stable or decreasing dose of corticosteroids for at least 5 days prior to baseline magnetic resonance imaging (MRI) or computed tomography (CT); if steroids are added or the steroids dose is increased between the date of the screening MRI or CT and the start of treatment, a new baseline MRI or CT is required
* Patients must be able to swallow whole capsules
* Ability to understand and the willingness to sign a written informed consent document
* For stage 2 GBM participants, a block of paraffin embedded tissue or 30 unstained slides at standard 4-5 um thickness from any prior surgery demonstrating GBM pathology must be available for submission
* Stage 2 endometrial and ovarian cancer patients must have at least one lesion amenable to biopsy; this determination will be made by a member of the interventional radiology team or surgical associate investigator and an associate investigator; this requirement is not necessary for patients in stage 1
* Solid tumor patients in stage 2 must have a diagnosis of papillary serous, endometrioid or clear cell endometrial carcinoma or, high grade serous, clear cell, endometrioid or mucinous ovarian, fallopian or primary peritoneal carcinoma

Exclusion Criteria:

* Concurrent administration of any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN0128 or bevacizumab
* For all stage 2 participants, no prior treatment with mTOR, PI3 kinase or Akt inhibitors; prior treatment with mTOR, PI3 kinase or Akt inhibitors allowed in stage 1 only
* For stage 2 GBM participants, no prior treatment with bevacizumab/vascular endothelial growth factor receptor (VEGFR) inhibitors; prior treatment with bevacizumab/VEGFR inhibitors is allowed in stage 1 for all participants, as well as stage 2 endometrial and ovarian cancer participants
* Stage 1 solid tumor and stage 2 endometrial and ovarian cancer participants with known central nervous system (CNS) metastatic lesions which are symptomatic and/or growing; patients previously treated for these conditions that are asymptomatic in the absence of corticosteroid therapy are allowed to enroll; brain metastasis must be stable for 1 month with verification by imaging (brain MRI completed at screening demonstrating no current evidence of progressive brain metastases); CNS imaging will not be mandated for asymptomatic patients with no history of CNS metastases
* Concurrent use of enzyme-inducing anti-epileptic drugs (EIAED); patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs; patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of MLN0128
* Subjects taking strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) and cytochrome P450, family 2, subfamily C, polypeptide 19 (CYP2C19) inhibitors and/or inducers should be considered with caution; alternative treatments that are less likely to affect MLN0128 metabolism, if available, should be considered; if a subject requires treatment with 1 or more of the strong CYP3A4 and CYP2C19 inhibitors and/or inducers, the principal investigator should be consulted
* Concurrent use of herbal supplements and other non-traditional medications; all herbal supplements and other non-traditional medications must be stopped before time of registration
* Concurrent use of anti-coagulants (warfarin, etc.) other than low-molecular weight heparin (LMWH); medication must be stopped before time of registration; if patient has recently been on anti-coagulants other than LMWH, patient must have international normalized ratio (INR) =< 2
* Evidence of any significant intracranial hemorrhage, as determined by the treating investigator, within 6 weeks from registration or as seen on most recent MRI prior to screening/baseline MRI
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* History of any of the following within 6 months prior to start of MLN0128:
* Left ventricular ejection fraction (LVEF) =< 55% as determined by multi gated acquisition (MUGA) scan or echocardiogram (ECHO)
* Heart failure >= New York Heart Association (NYHA) grade 3
* Significant ST depression of >= 1.5 mm in 2 or more leads and/or T wave inversions in >= 2 leads
* Complete left bundle branch block
* Right bundle branch block + left anterior hemiblock (bi-fascicular block)
* Congenital long QT syndrome
* QT interval corrected by Fridericia's formula (QTcF) > 450 msec on screening electrocardiogram (ECG)
* Requirement of inotropic support (excluding digoxin)
* History or presence of clinically significant ventricular or atrial tachyarrhythmias, or cardiac arrest
* Clinically significant resting bradycardia
* Presence of unstable atrial fibrillation (ventricular response > 100 beats per minute)
* Patients with stable atrial fibrillation are allowed in the study provided they do not meet the other cardiac exclusion criteria
* History of arrhythmia requiring an implantable cardiac defibrillator
* Angina pectoris =< 12 months prior to starting drug
* Acute myocardial infarction =< 12 months prior to starting drug
* Any valve disease Common Terminology Criteria for Adverse Events (CTCAE) grade
* Ischemic myocardial event including angina requiring therapy and artery revascularization procedures
* Placement of a pacemaker for control of rhythm
* Pulmonary embolism
* Ischemic cerebrovascular event, including transient ischemic attack (TIA) and artery revascularization procedures
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral MLN0128 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection that requires nutritional support)
* Use of hematopoietic colony-stimulating growth factors (e.g. filgrastim [G-CSF], sargramostim [GMCSF], lanimostim [M-CSF]) =< 2 weeks prior to starting study drug; erythropoietin, darbepoetin and erythropoietin-biosimilars are allowed for as long as they have been initiated at least 2 weeks prior to study enrollment
* Pregnant or nursing women; breastfeeding should be discontinued if the mother is treated with MLN0128
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; if an HIV-positive patient has adequate cluster of differentiation (CD4) counts (CD4 above the lower limit of institutional normal) and is on antiretroviral therapy with newer agents, which are not strong cytochrome (CYP) inhibitors, they will be eligible
* Uncontrolled high blood pressure (i.e., systolic blood pressure >= 160 mmHg, diastolic blood pressure >= 90 mmHg)
* Pulmonary hypertension
* Uncontrolled asthma or oxygen (O2) saturation < 90% by ABG (arterial blood gas) analysis or pulse oximetry on room air
* Participants with poorly controlled diabetes mellitus (defined as hemoglobin A1c [HbA1c] > 7%); subjects with a history of transient glucose intolerance due to corticosteroid administration are allowed in this study if all other inclusion/exclusion criteria are met
* Urine protein should be screened by urinalysis; if protein is 2+ or higher, 24 hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment
* Serious or non-healing wound, ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 1
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to day 1 therapy
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy within 7 days prior to day 1 therapy
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1
* Evidence of bleeding diathesis or coagulopathy
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2026-10-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Nayak, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 - Dose Level 1: Stage 1 (Dose Finding/Escalation Stage) - Dose Level 1:
  * 3 mg MLN0128 daily
  * + 10 mg/kg bevacizumab every 2 weeks
- Stage 1 - Dose Level 2: Stage 1 (Dose Finding/Escalation Stage) - Dose Level 2:
  * 4 mg MLN0128 daily
  * + 10 mg/kg bevacizumab every 2 weeks
- Stage 1 - Dose Level 3: Stage 1 (Dose Finding/Escalation Stage) - Dose Level 3:
  * 5 mg MLN0128 daily
  * + 10 mg/kg bevacizumab every 2 weeks
- Stage 2 - Maximum Tolerated Dose (MTD): Stage 2 - Expansion Cohort at Dose Level 3 - the Maximum Tolerated Dose (MTD) / Recommended Phase 2 Dose (RP2D):
  * 5 mg MLN0128 daily
  * + 10 mg/kg bevacizumab every 2 weeks
Period: Registration to Initiation of Therapy
Arm/Group | Stage 1 - Dose Level 1 | Stage 1 - Dose Level 2 | Stage 1 - Dose Level 3 | Stage 2 - Maximum Tolerated Dose (MTD)
Started | 3 | 3 | 6 | 38
Completed | 3 | 3 | 6 | 37
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Study Therapy
Arm/Group | Stage 1 - Dose Level 1 | Stage 1 - Dose Level 2 | Stage 1 - Dose Level 3 | Stage 2 - Maximum Tolerated Dose (MTD)
Started | 3 | 3 | 6 | 37
Completed | 3 | 3 | 6 | 37
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: 3 mg/day MLN0128
- Dose Level 2: 4 mg/day MLN0128
- Dose Level 3 (MTD): 5 mg/day MLN0128
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 (MTD) | Total
Number analyzed (Participants) | 3 | 3 | 43 | 49
Age, Continuous [Median (Full Range); unit: years] | 56 [55 to 65] | 42 [30 to 62] | 59 [36 to 84] | 59 [30 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 35 | 38
  Male | 2 | 1 | 8 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — National Institutes of Health (NIH) / Office of Management and Budget (OMB) Standards
  Participants
    Hispanic or Latino | 0 | 0 | 1 | 1
    Not Hispanic or Latino | 3 | 3 | 41 | 47
    Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — National Institutes of Health (NIH) / Office of Management and Budget (OMB) Standards
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 1 | 1
    White | 3 | 2 | 39 | 44
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 2 | 2
Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status [Median (Full Range); unit: units on a scale] — ECOG 0 = Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  ECOG 1 = Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  NOTE: Performance Status (PS) for patients with endometrial and ovarian cancer is reported via ECOG scale (0-5); PS for patients with glioblastoma is reported via Karnofsky (KPS) scale (100-0). Baseline PS for GBM patients has been converted from KPS to ECOG scale for reporting consistency.
  units on a scale | 0 [0 to 0] | 0 [0 to 1] | 1 [0 to 1] | 1 [0 to 1]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (R2PD) of Daily Oral MLN0128 When Administered With Bevacizumab
Description: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (R2PD) of TORC1/2 inhibitor MLN0128, determined according to incidence of dose-limiting toxicity, as graded using the National Cancer Institute (NCI) CTCAE version 4.0
Time Frame: 28 days
Measure: Number; unit: mg/day
Groups:
- Stage 1: Dose Escalation to Estimate MTD/RP2D: Participants enrolled onto Stage 1 - Dose escalation to estimate MTD/RP2D
Arm/Group | Stage 1: Dose Escalation to Estimate MTD/RP2D
Number analyzed (Participants) | 12
mg/day | 5

2. Primary Outcome: Most Common Related Toxicities That Led to Dose Hold/Reductions
Description: Most common related toxicities that led to dose hold/reductions (AEs graded according to NCI CTCAE version 4.0). Safety assessed through summaries of adverse events, changes in selected laboratory test results, changes in vital signs, and TORC1/2 inhibitor MLN0128 and bevacizumab exposure.
Time Frame: Up to 2 years
Population: AEs on the study are reported by dose level.
Measure: Number; unit: participants
Groups:
- Dose Level 1 - 3 mg MLN0128 Daily: Stage 1 - Dose Level 1 participants:
  * 3 mg MLN0128 daily
  * + 10 mg/kg bevacizumab every 2 weeks
- Dose Level 2 - 4 mg MLN0128 Daily: Stage 1 - Dose Level 2 participants:
  * 4 mg MLN0128 daily
  * + 10 mg/kg bevacizumab every 2 weeks
- Dose Level 3 - 5 mg MLN0128 Daily: Inclusive of both Stage 1 - Dose Level 3 participants and Stage 2 participants treated at the MTD:
  * 5 mg MLN0128 daily
  * + 10 mg/kg bevacizumab every 2 weeks
Arm/Group | Dose Level 1 - 3 mg MLN0128 Daily | Dose Level 2 - 4 mg MLN0128 Daily | Dose Level 3 - 5 mg MLN0128 Daily
Number analyzed (Participants) | 3 | 3 | 43
participants
  Grade 3 Altered mental status | 0 | 0 | 2
  Grade 3 Colon obstruction | 0 | 0 | 1
  Grade 3 Diarrhea | 0 | 0 | 1
  Grade 3 Fatigue | 0 | 0 | 3
  Grade 3 Hypercholesterolemia | 0 | 1 | 2
  Grade 3 Hypokalemia | 0 | 0 | 2
  Grade 3 Hypophosphatemia | 0 | 0 | 1
  Grade 3 Lymphopenia | 0 | 0 | 1
  Grade 3 Oral mucositis | 0 | 0 | 5
  Grade 3 Pruritus | 0 | 1 | 3
  Grade 3 Rash | 0 | 0 | 10
  Grade 3 Thrombocytopenia | 0 | 0 | 1
  Grade 3 Vomiting | 0 | 0 | 1
  Grade 1/2 Abdominal pain | 0 | 0 | 2
  Grade 1/2 Acute kidney injury | 0 | 0 | 2
  Grade 1/2 Anorexia | 0 | 0 | 2
  Grade 1/2 Constipation | 0 | 0 | 2
  Grade 1/2 Dehydration | 0 | 0 | 3
  Grade 1/2 Diarrhea | 0 | 1 | 5
  Grade 1/2 Fatigue | 0 | 0 | 8
  Grade 1/2 Fever | 0 | 0 | 1
  Grade 1/2 Hyperglycemia | 0 | 0 | 1
  Grade 1/2 Hypertriglyceridemia | 0 | 1 | 1
  Grade 1/2 Lymphopenia | 0 | 0 | 1
  Grade 1/2 Nausea | 0 | 0 | 3
  Grade 1/2 Oral mucositis | 0 | 0 | 4
  Grade 1/2 Pruritis | 0 | 0 | 6
  Grade 1/2 Pulmonary emboli | 0 | 0 | 1
  Grade 1/2 Rash | 0 | 1 | 11
  Grade 1/2 Thrombocytopenia | 0 | 0 | 6
  Grade 1/2 Vomiting | 1 | 0 | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined as follows:
  1. Non-GBM Solid Tumors (Endometrial & Ovarian Cancers) - using Response Evaluation Criteria In Solid Tumors Criteria (RECIST) guideline (v.1.1):
     * Target Lesions: >/= 20% increase in the sum of the longest diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
     * Non-Target Lesions: The appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
  2. GBM - Using the Response Assessment in Neuro-Oncology (RANO) criteria, any of the criteria below qualify for progression:
     * >/= 25% increase in sum of the products of perpendicular diameters of enhancing lesions on stable/increasing dose of corticosteroids
       * Significant increase in T2/FLAIR non-enhancing lesion on stable/increasing dose of corticosteroids
       * Any new lesion
       * Clear clinical deterioration not attributable to other cause
Time Frame: Up to 2 years
Population: * Given the limited sample sizes for Dose Levels 1 & 2 (3 patients each), the #s presented here may not be statistically valid.
  * Censoring & Final PFS #s: 9 patients treated @ Dose Level 3 were censored from PFS analysis for initiation of new therapy or withdrawal of consent. 2 additional patients treated at Dose Level 3 were censored from PFS analysis because they never had a useable scan on study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 (MTD)
Number analyzed (Participants) | 3 | 3 | 33
months | 1.6 [1.0 to NA] — Sample size of 3 patients is too low. | 7.3 [2.1 to NA] — Sample size of 3 patients is too low. | 5.4 [2.8 to 7.4]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR), defined as a Complete Response (CR) or Partial Response (PR) utilizing:
  1. RECIST criteria v.1.1 (Endometrial & Ovarian Cancers):
     * CR: Disappearance of all target & non-target lesions (+ normalization of tumor marker level)
     * PR: >/= 30% decrease in sum of the longest diameters of target lesions (from baseline) & no new lesions
  2. RANO criteria (GBM patients):
     * CR:
       * Disappearance of all enhancing measurable & non-measurable disease (sustained >/= 4 wks)
       * No new lesions
       * No steroids (physiologic replacement doses only)
       * Stable or improved non-enhancing lesions
       * Clinically stable or improved
     * PR:
       * >/= 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions (sustained >/= 4 wks)
       * No progression of non-measurable disease
       * No new lesions
       * Steroid </= dose at time of baseline scan
       * Stable or improved non-enhancing lesions
       * Clinically stable or improved
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: 3 mg MLN0128 Daily
- Dose Level 2: 4 mg MLN0128 Daily
- Dose Level 3 (MTD): 5 mg MLN0128 Daily
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 (MTD)
Number analyzed (Participants) | 3 | 3 | 43
Participants
  Complete Response | 1 | 0 | 0
  Partial Response | 0 | 0 | 8
  Stable Disease | 0 | 2 | 20
  Progressive Disease | 2 | 1 | 7
  Unevaluable | 0 | 0 | 8

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) listed for all patients by dose level.
Time Frame: Up to 4 years
Population: * Given the limited sample sizes for Dose Levels 1 & 2 (3 & 2 patients respectively), the #s presented here may not be statistically valid.
  * Censoring & Final OS #s: 1 patient treated at Dose Level 2 and 6 patients treated at Dose Level 3 were censored from OS analysis for withdrawal of consent or lost to follow-up, and were not followed for survival to their death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 (MTD)
Number analyzed (Participants) | 3 | 2 | 36
months | 7.9 [2.0 to NA] — Sample size of 3 patients is too small. | 11.6 [3.7 to NA] — Sample size of 2 patients is too small. | 9.3 [6.0 to 13.5]

6. Secondary Outcome: Number of Participants With Toxicities Leading to Missed Doses or Delays
Description: Number of Participants with Toxicities Leading to Missed Doses or Delays
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Dose Level 1 - 3 mg MLN0128 Daily | Dose Level 2 - 4 mg MLN0128 Daily | Dose Level 3 - 5 mg MLN0128 Daily
Number analyzed (Participants) | 3 | 3 | 43
participants | 1 | 1 | 33

7. Secondary Outcome: Number of Participants Who Had an MLN0128 Dose-Reduction On Study
Description: Number of patients who had to have their MLN0128 dose reduced while on study.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 3 mg MLN0128 Daily | Dose Level 2 - 4 mg MLN0128 Daily | Dose Level 3 - 5 mg MLN0128 Daily
Number analyzed (Participants) | 3 | 3 | 43
Participants | 0 | 2 | 24

8. Secondary Outcome: Number of Patients That Discontinue Study Drugs Due to Treatment Related Toxicity
Description: Number of patients that discontinue study drugs due to treatment related toxicity; percentage will be summarized.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 3 mg MLN0128 Daily | Dose Level 2 - 4 mg MLN0128 Daily | Dose Level 3 - 5 mg MLN0128 Daily
Number analyzed (Participants) | 3 | 3 | 43
Participants | 0 | 0 | 10

9. Other Pre Specified Outcome: Cerebrospinal Fluid (CSF) Penetration of TORC1/2 Inhibitor MLN0128, Evaluated Using Plasma and CSF Pharmacokinetic (PK) Parameters of MLN0128
Description: Plasma and CSF PK levels of TORC1/2 inhibitor MLN0128 obtained before and after bevacizumab administration will be evaluated and summarized. The ration of plasma to CSF PK levels will also be summarized.
Time Frame: 2-3 hours post-dose day 15 of course 1 and day 1 of course 2
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Markers Associated With Dysregulated Cell Signaling
Description: The biomarkers predicting response to mechanistic target of rapamycin (mTOR) inhibitor activity will be resulted by dose level and response status.
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Phosphorylated Proteins Within Tumor Biopsies From Patients With Ovarian and Endometrial Cancers
Time Frame: Baseline to within 7 days after last study drug or within 7 days after decision to end treatment
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Circulating Plasma Levels of Angiogenic Growth Factors in Patients With Ovarian and Endometrial Cancers
Time Frame: Baseline to day 1 of last course of treatment
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Mutation Analysis of Tissue From Biopsies of Patients With Ovarian and Endometrial Cancers
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse Events monitored/assessed up to 2 years and All-Cause Mortality was monitored until death, withdrawal of consent, or lost-to-follow-up (maximum # of days a patient was on study was 1443 days).
Arm/Group | Dose Level 1 - 3 mg MLN0128 Daily | Dose Level 2 - 4 mg MLN0128 Daily | Dose Level 3 - 5 mg MLN0128 Daily
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 36/43
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 19/43
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 - 3 mg MLN0128 Daily (N=3) | Dose Level 2 - 4 mg MLN0128 Daily (N=3) | Dose Level 3 - 5 mg MLN0128 Daily (N=43)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 4
Fever (General disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 3
Death NOS (General disorders) | 0 | 0 | 2
Dysphasia (Nervous system disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 4
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Other, specify: Death due to progression of endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Other, specify - mood alteration (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 - 3 mg MLN0128 Daily (N=3) | Dose Level 2 - 4 mg MLN0128 Daily (N=3) | Dose Level 3 - 5 mg MLN0128 Daily (N=43)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 9
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 7
Constipation (Gastrointestinal disorders) | 0 | 1 | 13
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 21
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 4
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 3
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 22
Nausea (Gastrointestinal disorders) | 3 | 1 | 22
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 12
Chills (General disorders) | 0 | 0 | 5
Edema face (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 0 | 0 | 9
Fatigue (General disorders) | 2 | 2 | 27
Fever (General disorders) | 0 | 0 | 3
Pain (General disorders) | 0 | 0 | 3
Skin infection (Infections and infestations) | 0 | 0 | 3
Tooth infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 10
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 7
Alanine aminotransferase increased (Investigations) | 0 | 0 | 9
Alkaline phosphatase increased (Investigations) | 0 | 0 | 11
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 11
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Cholesterol high (Investigations) | 1 | 1 | 16
Creatinine increased (Investigations) | 0 | 1 | 13
Other, specify: LDH Increased (Investigations) | 0 | 0 | 8
Lymphocyte count decreased (Investigations) | 0 | 1 | 16
Neutrophil count decreased (Investigations) | 0 | 0 | 4
Platelet count decreased (Investigations) | 0 | 1 | 21
Weight loss (Investigations) | 0 | 0 | 13
White blood cell decreased (Investigations) | 0 | 0 | 11
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 21
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 25
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 9
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 7
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 4
Dizziness (Nervous system disorders) | 1 | 0 | 5
Dysgeusia (Nervous system disorders) | 0 | 1 | 10
Headache (Nervous system disorders) | 1 | 1 | 8
Memory impairment (Nervous system disorders) | 0 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 4
Sinus pain (Nervous system disorders) | 0 | 0 | 3
Tremor (Nervous system disorders) | 0 | 0 | 11
Anxiety (Psychiatric disorders) | 0 | 0 | 4
Confusion (Psychiatric disorders) | 0 | 1 | 6
Depression (Psychiatric disorders) | 0 | 0 | 9
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 14
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 10
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 25
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 18
Hypertension (Vascular disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 4
Paronychia (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Investigations - Other, specify: Globus sensation (Investigations) | 1 | 0 | 0
Ear and labyrinth disorders - Other, specify: Ears bothering with mild fluid build-up (Ear and labyrinth disorders) | 0 | 1 | 0
Eye disorders - Other, specify: Decrease in vision (Eye disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT02142803/Prot_SAP_000.pdf